CLINICAL TRIAL: NCT00786669
Title: A Pilot Study of the Addition of Bevacizumab to Vincristine, Oral Irinotecan, and Temozolomide (VOIT Regimen) for Relapsed/Refractory Pediatric Solid Tumors
Brief Title: A Pilot Study of the Addition of Bevacizumab to VOIT Regimen for Relapsed/Refractory Pediatric Solid Tumors
Acronym: VITAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VITAC
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2015-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Bevacizumab; Temozolomide; Vincristine; Irinotecan; Cefixime; Cefpodoxime Proxetil; Cefpodoxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab+TEM/VCR/IRN/CEF (Experimental): Bevacizumab(IV) 15 mg/Kg on day 1 every 3 weeks for up to 6 cycles
  Temozolomide (TEM) 100 mg/m2/day po on Days 1-5 every 3 weeks for up to 6 cycles. For patients under 0.5 m2 BSA, TEM = 3.3 mg/kg/day po on Days 1-5.
  Vincristine (VCR) 1.5 mg/m2 on Day 1 (max dose 2 mg) administered as an IV bolus every 3 weeks for up to 6 cycles. For patients <0.5 m2 BSA, VCR dose = 0.05 mg/kg (maximum dose 2 mg).
  Irinotecan (IRN) 90 mg/m2/day po on Days 1-5 every 3 weeks for up to 6 cycles
  Cefexime (CEF) 8 mg/kg/day (max. daily dose 400 mg) of cefixime or 5 mg/kg/dose bid (max. daily dose 400 mg) of cefpodoxime starting Day -1 BEFORE chemotherapy and continuing EVERY DAY while on study, or for 2 days after last dose of chemotherapy if treatment stopped early for disease progression or toxicity
  Interventions: Drug: Bevacizumab; Drug: Temozolomide; Drug: Vincristine; Drug: Irinotecan; Drug: Cefixime

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (IV) 15 mg/Kg on day 1 every 3 weeks for up to 6 cycles
  Other Names: rhuMAb VEGF; Avastin
Drug: Temozolomide — 100 mg/m2/day po on Days 1-5 every 3 weeks for up to 6 cycles. For patients under 0.5 m2 BSA, TEM = 3.3 mg/kg/day po on Days 1-5.
  Other Names: Temodar; TEM
Drug: Vincristine — 1.5 mg/m2 on Day 1 (max dose 2 mg) administered as an IV bolus every 3 weeks for up to 6 cycles. For patients <0.5 m2 BSA, VCR dose = 0.05 mg/kg (maximum dose 2 mg).
  Other Names: VCR; Oncovin
Drug: Irinotecan — 90 mg/m2/day po on Days 1-5 every 3 weeks for up to 6 cycles
  Other Names: CPT-11; Camptothecin-11; Camptosar®; IRN
Drug: Cefixime — 8 mg/kg/day (max. daily dose 400 mg) of cefixime or 5 mg/kg/dose bid (max. daily dose 400 mg) of cefpodoxime starting Day -1 BEFORE chemotherapy and continuing EVERY DAY while on study, or for 2 days after last dose of chemotherapy if treatment stopped early for disease progression or toxicity
  Other Names: Suprax®; Vantin®; Cefpodoxime; CEF

SUMMARY:
The purpose of this research study is to test the safety and of adding bevacizumab to the established regimen of vincristine, oral irinotecan, and temozolomide (VOIT) and see what effects it has in pediatric patients with relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
A recent Children's Oncology Group study evaluated the 3-drug combination of vincristine, oral irinotecan, and temozolomide (VOIT), and found it to be safe and tolerable in pediatric patients. This VOIT regimen may be useful for a variety of childhood cancers.

Additional data suggests that the beneficial effects of irinotecan can be improved by giving it with bevacizumab. Bevacizumab is a monoclonal antibody that works against a protein called "vascular endothelial growth factor" (VEGF). In cancer treatment, it is used to reduce tumor growth by blocking the formation of new blood vessels.

All of the drugs used in this study have been approved by the Food and Drug Administration (FDA) for use in adults with certain cancer types. However, the combination of drugs in this study is considered experimental because the FDA has not approved them to be used together.

Each drug has been given by itself to children before, and the combination of temozolomide, irinotecan, and vincristine has been given to children in more than one clinical trial. This is the first study in which all four of the drugs (vincristine, oral irinotecan, temozolomide, and bevacizumab) will be given together to children.

Up to 20 pediatric patients will receive therapy. The previously established bevacizumab dose of 15 mg/kg will be administered by intravenous infusion on day 1 at the start of every 3-week course. Intravenous vincristine will be given on day 1, oral irinotecan on days 1-5, and oral temozolomide on days 1-5. Courses will be repeated as frequently as every three weeks in patients who do not have evidence of disease progression and who have adequate recovery from previous courses. Cephalosporin antibiotics will be used to reduce irinotecan-associated diarrhea.

Patients will be monitored on the study for toxicity and response for up to 6 courses.

ELIGIBILITY:
Inclusion Criteria:

* Between 1 and 30 years of age, inclusive, at the time of study entry
* Histologic verification of a solid tumor or CNS tumor at either original diagnosis or relapse. Exceptions to the requirement for biopsy include patients with primary brainstem or optic pathway tumors.
* Current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Karnofsky ≥ 50% for patients > 10 years of age and Lansky ≥ 50 for patients < 10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score. Life expectancy must be ≥ 8 weeks.
* Agreement to use an effective contraception method during and for 30 days after treatment.
* Prior treatment with vincristine, temozolomide, or irinotecan is allowed, although patients must not have had disease progression while receiving either irinotecan or temozolomide. Prior treatment with bevacizumab is not allowed.
* Adequate Bone Marrow (Peripheral ANC ≥ 750/uL, PLT ≥ 75,000/uL transfusion independent, Hgb ≥ 8.0 gm/dL), renal (negative urine dipstick for protein, OR < 1000 mg protein/24-hour urine collection, Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2), and liver function (Bilirubin ≤ 1.5 ULN, SGPT ≤ 5 ULN, Serum albumin ≥ 2 g/dL).
* Adequate blood clotting (INR, Fibrinogen, and PTT < grade 2).

Exclusion Criteria:

* Concomitant Medications: Growth factors that support platelet or white cell number or function administered within the past 3 days, currently receiving investigational drugs, or who have received an investigational drug within the last 7 days, currently receiving other anti-cancer agents, currently taking phenobarbital, phenytoin, carbamazepine, oxcarbazepine (Trileptal), rifampin, voriconazole, itraconazole, ketoconazole or other systemically-administered azole antifungal drugs, aprepitant (Emend), or St. John's Wort, requiring antihypertensive agents at the time of enrollment, receiving medications known to inhibit platelet function or known to selectively inhibit cyclooxygenase activity, with the exception of acetaminophen.
* Require IV antibiotics at time of enrollment, or who are currently receiving treatment for Clostridium difficile infection.
* Must not have been previously diagnosed with a deep venous or arterial thrombosis (including pulmonary embolism), and must not have a known thrombophilic condition.
* Experienced arterial thromboembolic events, including transient ischemic attacks or cerebrovascular accidents, within the last year. Must not have a history of myocardial infarction, severe or unstable angina, or clinically significant peripheral vascular disease.
* Documented, chronic non-healing wound, ulcer, or bone fracture, as well as patients who have had a major surgical procedure or significant traumatic injury within 28 days prior to beginning therapy.
* Recent (within last 6 months) hemoptysis (≥ ½ teaspoon of red blood).

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Toxicities of adding bevacizumab to the established VOIT regimen using cefixime to reduce irinotecan-associated diarrhea. | During treatment course
  Define the toxicities of adding bevacizumab to the established vincristine, oral irinotecan, and temozolomide (VOIT) regimen using cefixime to reduce irinotecan-associated diarrhea.

SECONDARY OUTCOMES:
Preliminarily definition of the antitumor activity of this drug combination within the confines of a small pilot trial. | Two years
  Preliminarily define the antitumor activity of this drug combination within the confines of a small pilot trial.
Feasibility assessment of the collection and analysis of serum DNA for methylation of the MGMT promotor. | Two years
  To assess the feasibility of collecting and analyzing serum Deoxyribonucleic acid (DNA) for methylation of the methylguanine-deoxyribonucleic acid methyltransferase (MGMT) promotor.
Comparison of free and total levels of VEGF in serum following treatment with bevacizumab. | Two Years
  Compare free and total levels of Vascular endothelial growth factor (VEGF) in serum following treatment with bevacizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Turpin, D.O., Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States